CLINICAL TRIAL: NCT04444180
Title: The Predictive Role of Self Representation in Transition of Individuals at Clinical High Risk for Psychosis -- a Study on the Clinical Application of Virtual Hand Illusion
Brief Title: The Predictive Role of Self-representation in Transition of Individuals at Clinical High Risk for Psychosis
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: CRC2018YB01
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Clinical High Risk for Psychosis
Keywords: sense of ownership; sense of agency; virtual hand illusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Clinical high risk for psychosis (CHR): No intervention. Just use virtual hand illusion (VHI) paradigm to observe the outcome of individuals with CHR at one-year follow-up node and analyze the predictive role of self-representation in transition into psychosis.
  Interventions: Diagnostic Test: Virtual hand illusion (VHI)
- First episode of schizophrenia (FES): In contrast to FES, it is anticipated to observe CHR individuals with similar behavioral performance to FES may presented higher risk of transition.
  Interventions: Diagnostic Test: Virtual hand illusion (VHI)
- Healthy control (HC): In contrast to HC, it is anticipated to observe CHR individuals with similar behavioral performance to HC may presented lower risk of transition.
  Interventions: Diagnostic Test: Virtual hand illusion (VHI)

INTERVENTIONS:
Diagnostic Test: Virtual hand illusion (VHI) — Using VHI, the two basic self-representation of sense of ownership and sense of agency of the subjects will be observed.

SUMMARY:
Schizophrenia is one of the most consumptive diseases, which brings great loss to patients and their families, and even to the society. Clinical High Risk for Psychosis (CHR) is a concept put forward on the basis of the prodromal stage of schizophrenia. Over the past 20 years, the identification and intervention of CHR has become the focus of psychiatric research, with the primary goal of early identification of biomarkers of susceptibility to schizophrenia and the development of individualized interventions to prevent or delay progression. Longitudinal studies have shown that CHR converted to schizophrenia mainly within two years, with a risk of about 30 percent. Self-disorder is one of the core characteristics of schizophrenia. The two most basic experiences of self-representation are sense of ownership and sense of agency. Sense of ownership refers to the sense that "I" perceives "my" body, while sense of agency refers to the sense that "I" experiences "my" actions and their consequences are initiated by "me". Some studies have shown that patients with schizophrenia show defects in the sense of ownership and agency. The most commonly used paradigm for observing "sense of ownership" and "sense of agency" is the rubber hand illusion (RHI) or the virtual hand illusion (VHI). In this study, the VHI experimental paradigm will be used to detect the self-representation of the individuals at high risk for psychosis, and the clinical outcome will be observed for one year.The hypothesis is that the subjects who exhibit abnormal illusion experience in VHI experiment are more likely to transition into psychotic disorders.

DETAILED DESCRIPTION:
This study is conducted according to the tenets of the Declaration of Helsinki. All participants are recruited at the Shanghai Mental Health Center (SMHC) or its affiliate, the Shanghai Psychotherapy and Psychological Counseling Center (SPCC) with written informed consent, approved by the Research Ethics Committee of SMHC. For those younger than 18 years, both the adolescents and their next of kin or legal guardians are provided informed consents. The outpatients are recommended by doctors to participate in our CHR screening. After being screened and interviewed, those who meet the inclusion criteria are informed and signed written informed consent. Once the subjects are recruited, clinical evaluation, VHI and MCCB test will be conducted. In addition, CHR individuals will be followed up at one-year node.

ELIGIBILITY:
Inclusion Criteria:

* For CHR individuals, meet the criteria of psychosis-risk syndromes after rating by structured interview for psychosis high risk syndrome.
* For FES patients, meet diagnostic criteria for schizophrenia in the DSM-IV.
* For HC individuals, gender composition, age range, educational level are matched with CHR individuals.
* Understand and sign written informed consent.

Exclusion Criteria:

* For CHR individuals, exclude individuals with other axis I or II mental disorders, which can explain the abnormal experience.
* For CHR and FES patients, exclude those patients taking antipsychotics for more than two weeks.
* For HC individuals, exclude those with family history of mental disorders
* With a history of substance dependence.
* Use of medications that may affect mental and cognitive functions.
* With central nervous system disorder, that cuase symptoms or interfere with judgment.
* Traumatic brain injury score is 7 or more.
* With serious or unstable physical diseases.
* With perceptual developmental disorders.
* IQ<70.

Ages: 11 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study mainly observe the behavioral representation and its predictive role in transition outcome of CHR individuals, who meeting the criteria of psychosis-risk syndromes (COPS) for the existence of one or more of psychosis high risk syndromes, such as brief intermittent psychotic syndrome (BIPS), attenuated positive symptom syndrome (APSS), and genetic risk and deterioration syndrome (DRDS).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Behavioral indicators | Baseline
  To compare the behavioral performance in VHI experimental paradigm among the three groups of CHR, FES, and HC
Predictive indicators | One-year follow-up node
  To analyze the predictive role of self-representation in transition of CHR into psychosis

SECONDARY OUTCOMES:
Resting-state brain functional connectivity (FC) | Baseline
  To observe the relationship of the behavioral performance in VHI experimental paradigm with the Resting-state brain functional connectivity
Event-related potential technique | Baseline
  To observe the relationship of the behavioral performance in VHI experimental paradigm with the error-related negativity
Neurocognitive function | Baseline
  To observe the relationship of the behavioral performance in VHI experimental paradigm with the neurocognitive functions
Other predictive indicators | One-year follow-up node
  To analyze the predictive role of FC and neurocognitive functions related to self-representation in transition of CHR into psychosis

CONTACTS AND LOCATIONS:
Overall Officials: Jijun Wang, Doctoral, Study Chair — Shanghai Mental Health Center; Tianhong Zhang, Doctoral, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Raballo A, Monducci E, Ferrara M, Fiori Nastro P, Dario C; RODIN group. Developmental vulnerability to psychosis: Selective aggregation of basic self-disturbance in early onset schizophrenia. Schizophr Res. 2018 Nov;201:367-372. doi: 10.1016/j.schres.2018.05.012. Epub 2018 May 25. PMID 29804931
- [Result] Ebisch SJH, Aleman A. The fragmented self: imbalance between intrinsic and extrinsic self-networks in psychotic disorders. Lancet Psychiatry. 2016 Aug;3(8):784-790. doi: 10.1016/S2215-0366(16)00045-6. Epub 2016 Jun 30. PMID 27374147
- [Result] Newen A, Vogeley K. Self-representation: searching for a neural signature of self-consciousness. Conscious Cogn. 2003 Dec;12(4):529-43. doi: 10.1016/s1053-8100(03)00080-1. PMID 14656496
- [Result] Synofzik M, Vosgerau G, Newen A. I move, therefore I am: a new theoretical framework to investigate agency and ownership. Conscious Cogn. 2008 Jun;17(2):411-24. doi: 10.1016/j.concog.2008.03.008. Epub 2008 Apr 14. PMID 18411059
- [Result] Shaqiri A, Roinishvili M, Kaliuzhna M, Favrod O, Chkonia E, Herzog MH, Blanke O, Salomon R. Rethinking Body Ownership in Schizophrenia: Experimental and Meta-analytical Approaches Show no Evidence for Deficits. Schizophr Bull. 2018 Apr 6;44(3):643-652. doi: 10.1093/schbul/sbx098. PMID 29036731
- [Result] Germine L, Benson TL, Cohen F, Hooker CI. Psychosis-proneness and the rubber hand illusion of body ownership. Psychiatry Res. 2013 May 15;207(1-2):45-52. doi: 10.1016/j.psychres.2012.11.022. Epub 2012 Dec 28. PMID 23273611
- [Result] Fusar-Poli P, Cappucciati M, Borgwardt S, Woods SW, Addington J, Nelson B, Nieman DH, Stahl DR, Rutigliano G, Riecher-Rossler A, Simon AE, Mizuno M, Lee TY, Kwon JS, Lam MM, Perez J, Keri S, Amminger P, Metzler S, Kawohl W, Rossler W, Lee J, Labad J, Ziermans T, An SK, Liu CC, Woodberry KA, Braham A, Corcoran C, McGorry P, Yung AR, McGuire PK. Heterogeneity of Psychosis Risk Within Individuals at Clinical High Risk: A Meta-analytical Stratification. JAMA Psychiatry. 2016 Feb;73(2):113-20. doi: 10.1001/jamapsychiatry.2015.2324. PMID 26719911